CLINICAL TRIAL: NCT05892289
Title: Feasibility and Safety of Robotic Assisted Proximal Gastrectomy With Double-flap Technique for Proximal Early Gastric Cancer: a Phase II, Multi-center, Single-arm Clinical Study
Brief Title: Feasibility and Safety of Robotic Assisted Proximal Gastrectomy With Double-flap Technique for Proximal Early Gastric Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Collaborators: First Affiliated Hospital of Guangxi Medical University (Other); First Affiliated Hospital of Kunming Medical University (Other); First Hospital of China Medical University (Other); Gansu Provincial Hospital (Other); Qilu Hospital of Shandong University (Other); Shandong Provincial Hospital (Other Government); Sichuan Cancer Hospital and Research Institute (Other); Sichuan Provincial People's Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); LanZhou University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Tianjin Medical University Cancer Institute and Hospital (Other); Zunyi Medical College (Other); Liaoning Cancer Hospital & Institute (Other); Qinghai Province Cancer Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2022-275-02
Record Dates: First submitted 2023-05-04; First posted 2023-06-07 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Stomach Neoplasms
Keywords: Robotic Surgical Procedures; minimally invasive surgical procedures; stomach neoplasm; Gastrectomy; Reflux Esophagitis
MeSH Terms: conditions — Stomach Neoplasms; Esophagitis, Peptic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Robotic assisted proximal gastrectomy with double-flap technique (Experimental)
  Interventions: Procedure: Robotic assisted proximal gastrectomy with double-flap technique

INTERVENTIONS:
Procedure: Robotic assisted proximal gastrectomy with double-flap technique — Patients in this group receive robotic assisted proximal gastrectomy with D1+/D2 lymph node dissection(D1+ for stage IA：Nos.1, 2, 3a, 4 sa, 4 sb, 7, 8a, 9，11p；D2 for stage IB: Nos.1, 2, 3a, 4 sa, 4 sb, 7, 8a, 9，11p and 11d).The double-flap technique is used for the digestive tract reconstruction.

SUMMARY:
Proximal early gastric cancer can choose radical total gastrectomy or proximal gastrectomy. The patients have poor nutritional status and quality of life after total gastrectomy. Compare to total gastrectomy, the nutritional status can improve after proximal gastrectomy . But if use simple esophagogastric anastomosis for proximal gastrectomy, the incidence of postoperative reflux esophagitis is high, which seriously affects the quality of life, and the short-term outcome is poorer than the total gastrectomy. If the incidence of postoperative reflux esophagitis can be reduced, proximal gastrectomy would be the treatment choice for proximal early gastric cancer, which may more improve both quality of life and nutritional condition than total gastrectomy.

Double-flap technique is a new surgical reconstruction procedure between esophagus and remnant stomach. It can reduce the occurrence of reflux oesophagitis through reconstruction a simulative cardia. At present, the technique has been carried out in some hospitals in China but still lack large-scale prospective studies and evidence of evidence-based medicine. At present, some retrospective studies have shown that robotic assisted proximal gastrectomy with double-flap technique is safe and effective, and the learning curve is shorter than laparoscopic surgery. The applicant have finished two robotic assisted proximal gastrectomy with double-flap technique cases. Two patients recovered well after surgery, with no occurrence of anastomotic leakage or stenosis and the postoperative quality of life was good. Now we plan to conduct a multi-center, single arm study on proximal early gastric cancer patients(T1N0-1M0 and T2N0M0) to evaluate the feasibility of robotic assisted proximal gastrectomy with double-flap technique , and to evaluate the surgical and oncological safety of this surgical method. Aim to provide initial evidence of evidence-based medicine for its clinical application..

ELIGIBILITY:
Inclusion Criteria:

1. 20 years ≤ age ≤ 80 years
2. The primary gastric lesions were located in the proximal third of the stomach
3. histologically proven gastric adenocarcinoma (by preoperative gastrofiberscopy)
4. clinical stage IA (T1N0M0) or IB (T1N1M0 / T2N0M0) according to the 8th edition of the American Joint Committee on Cancer System(Clinical stage was determined based on the finding of endoscopic ultrasonography and/or thoraco-abdominal contrast-enhanced computed tomography)
5. scheduled for robotic assisted proximal gastrectomy with D1+/D2 lymphadenectomy, and possible for R0 surgery by this procedures (Lymphadenectomy is performed on the basis of the criteria of the Japanese Gastric Cancer Treatment Guidelines 2021 (6th edition).).
6. The preoperative American Society of Anesthesiologists (ASA) physical status was I-III;
7. The patient's cardiopulmonary function can tolerate robotic assisted surgery;
8. The subjects have signed the informed consent form.

Exclusion Criteria:

1. history of upper abdominal surgery and not suitable for robotic assisted surgery
2. the tumor invades the esophagus 3cm above gastro-esophageal junction (Z-line)
3. with other malignant diseases or have suffered from other malignant diseases within 5 years
4. Excessive tension for esophagogastric anastomosis and require changing the reconstruction procedure
5. women are pregnant or in lactation period
6. Suffering from serious mental illness
7. history of continuous systemic corticosteroid or immunosuppressive drug treatment within 1 month

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2026-12-10 (Estimated); Study Completion 2026-12-10 (Estimated)

PRIMARY OUTCOMES:
The Proportion of Patients With Reflux Esophagitis Within 12 Months Postoperatively | 12 months postoperatively
  During follow-up endoscopy 1 year after surgery, reflux esophagitis were graded according to the Los Angeles (LA) classification.

SECONDARY OUTCOMES:
Quality of Life after Surgery | Follow-up evaluations are performed 3, 6 and 12 months postoperatively
  Quality of life(QoL) is evaluated using the European Organization for Research and Treatment of Cancer (EORTC) 30-item core QoL (QLQ-C30 ver.3.0). Higher scores mean a worse outcome.
Gastrointestinal Symptoms after Surgery | Follow-up evaluations are performed 3, 6 and 12 months postoperatively
  gastrointestinal symptoms are assessed by Gastrointestinal Quality of Life Index (GIQLI) questionnaires. Higher scores mean a better outcome.
Changes in total protein at Follow-up | Follow-up evaluations are performed 3, 6 and 12 months postoperatively.
  blood total protein(g/L) levels
Changes in serum albumin at Follow-up | Follow-up evaluations are performed 3, 6 and 12 months postoperatively.
  blood serum albumin(g/L) levels
Changes in prealbumin at Follow-up | Follow-up evaluations are performed 3, 6 and 12 months postoperatively.
  blood prealbumin(g/L) levels
Changes in hemoglobin at Follow-up | Follow-up evaluations are performed 3, 6 and 12 months postoperatively.
  blood hemoglobin(g/L) levels
Changes in Vitamin B12 at Follow-up | Follow-up evaluations are performed 3, 6 and 12 months postoperatively.
  blood Vitamin B12(μg/ml) levels
Late Postoperative Morbidity | Follow-up evaluations are performed 3, 6 and 12 months postoperatively.
  adhesive ileus, anastomosis stenosis, malnutrition, dumping syndrome. All postoperative complications are classified according to the Clavien-Dindo(CD) classification standard.
Early Postoperative Morbidity | From surgery to discharge, up to 30 days
  operation wound with seroma, hematoma, infection, dehiscence, or evisceration, anastomotic leakage, anastomotic bleeding, abdominal bleeding, abdominal abscess, intestinal obstruction morbidity, gastrointestinal bleeding, gastroparesis, postoperative pancreatitis, pancreatic fistula, chylous leakage, lung morbidity, cerebrovascular morbidity, cardiovascular morbidity, deep vein thrombosis, cholecystitis, liver dysfunction, kidney dysfunction. All postoperative complications are classified according to the Clavien-Dindo(CD) classification standard.
Short-term Clinical Outcome After Surgery | From surgery to discharge, up to 30 days
  time to pass gas(hours)
Short-term Clinical Outcome After Surgery | From surgery to discharge, up to 30 days
  time to oral intake(hours)
Short-term Clinical Outcome After Surgery | From surgery to discharge, up to 30 days
  time to indwell gastric tube(hours)
Short-term Clinical Outcome After Surgery | From surgery to discharge, up to 30 days
  length of postoperative hospitalisation(days)
Surgical Characteristics | 24 hours postoperatively
  operative time(minutes)
Surgical Characteristics | 24 hours postoperatively
  time for reconstruction the digestive tract(minutes) during surgery
Surgical Characteristics | 24 hours postoperatively
  blood loss during surgery(ml)
Quality of Life postoperatively | Follow-up evaluations are performed 3, 6 and 12 months postoperatively
  Quality of life(QoL) is evaluated using the European Organization for Research and Treatment of Cancer (EORTC) gastric cancer module (QLQ-STO22) questionnaire. Higher scores mean a worse outcome.
Pathological Characteristics | 1 week postoperatively
  R0 resection rate. R0 resection represents complete resection of the tumor, meaning there is no residual tumor.
Pathological Characteristics | 1 week postoperatively
  lymph nodes dissection extent for each patient in the surgery
Pathological Characteristics | 1 week postoperatively
  number of dissected lymph nodes for each patient in the surgery
body mass index postoperatively | Follow-up evaluations are performed 3, 6 and 12 months postoperatively.
  body mass index(kg/m^2)
pain assessment postoperatively | Day 1 postoperatively
  We measured the pain score using visual analog scale(VAS) at 24 h after the surgery is completed. Higher scores mean a worse outcome.
Proportion of participants die after surgery | From surgery to discharge, up to 30 days
  mortality rate
Proportion of participants need to rehospitalized after surgery | From surgery to discharge, up to 30 days
  rehospitalization rate

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
The data sets generated and/or analysed during the current study are not publicly available due to governmental policy regarding individual information. However, they are available from the Sun Yat-Sen Memorial Hospital data center upon reasonable request, subject to approval by the Sun Yat-Sen Memorial Hospital Ethics Committee and the Data and Safety Monitoring Committee. This will be after the publication of the main findings, in line with standard data-sharing practices for clinical trial data sets. The Sun Yat-Sen Memorial Hospital data center will ensure the confidentiality of all participants' data and will not disclose information by which participants may be identified to any third party other than those directly involved in the treatment of the participant and organisations for which the participant has provided explicit consent for data transfer.

REFERENCES:
- [Derived] Zhong G, Xie Y, Chen G, Zhu Y, Yang B, Tan J, Han F, Zhou S. Assessing the feasibility and safety of robotic-assisted proximal gastrectomy with double-flap technique for proximal early gastric cancer: study protocol for a phase II, multicentre, single-arm clinical trial. BMJ Open. 2025 Aug 10;15(8):e094661. doi: 10.1136/bmjopen-2024-094661. PMID 40789587